CLINICAL TRIAL: NCT02398929
Title: An Open Label, Pharmacogenetic Study of Bisoprolol Treatment in Patients With Uncontrolled Essential Hypertension (BRAVE)
Brief Title: BRAVE Study With Uncontrolled Essential Hypertension (BRAVE Study)
Acronym: BRAVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Brian Tomlinson, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 200 006 621
Record Dates: First submitted 2015-03-17; First posted 2015-03-26 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bisoprolol 2.5 mg (Other): Bisoprolol 2.5 mg will be given once daily following run-in placebo for 2 weeks
  Interventions: Drug: Bisoprolol 2.5 mg; Drug: Placebo

INTERVENTIONS:
Drug: Bisoprolol 2.5 mg — Bisoprolol 2.5 mg will be given once daily
  Other Names: Concor
Drug: Placebo — Placebo tablets will be given once daily for 2 weeks during the run-in period.
  Other Names: Run-in

SUMMARY:
This is an open-label, placebo run-in study to investigate the genetic and biomedical predictors of blood pressure response to bisoprolol. After informed consent is obtained, subjects will be withdrawn from previous antihypertensive therapy and given placebo for at least 2 weeks. Compliance will be assessed using pill counting, and any subject will a compliance less than 80% during the placebo run-in period will be excluded from the study. Bisoprolol 2.5 mg will be given once daily for 6 weeks. At baseline and after 6 weeks on bisoprolol 2.5 mg the clinic sitting blood pressure, 24-hour ambulatory blood pressure (if the patient is willing to do this), clinical characteristics and biochemical profile will be measured. Central aortic blood pressure will be measured with the A-PULSE device at baseline and after 6 weeks treatment.

After completing 6 weeks treatment with bisoprolol 2.5 mg daily, the patient will continue treatment with bisoprolol for a total of 24 weeks unless there is any adverse event that requires discontinuation of bisoprolol.

DETAILED DESCRIPTION:
Patients with uncontrolled essential hypertension aged 18-79 years on no antihypertensive treatment with sitting clinic systolic blood pressure of 140-169 mmHg and/or a sitting clinic diastolic blood pressure of 90-109 mmHg, or for patients with diabetes mellitus or with chronic kidney disease with sitting clinic systolic blood pressure of 130-169 mmHg and / or a sitting clinic diastolic blood pressure of 80-109 mmHg and heart rate > 70 at baseline (before starting bisoprolol treatment) will be enrolled. Patients on other antihypertensive treatments who are experiencing side effects or whose blood pressure may not be well controlled can also enter if they can continue on a stable dose of a calcium channel blocker, either amlodipine or nifedipine retard throughout the study.

Patients will be treated with bisoprolol 2.5mg daily for a total of 26 weeks. The primary endpoint will be the influence of common genetic polymorphisms on clinic sitting blood pressure or ambulatory blood pressure (ABP) response to bisoprolol 2.5 mg after 6 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential hypertension
* For uncomplicated hypertensive patients on no antihypertensive treatment, sitting clinic systolic blood pressure of 140-169 mmHg and / or a sitting clinic diastolic blood pressure of 90-109 mmHg.
* For patients with diabetes mellitus or with chronic kidney disease, sitting clinic systolic blood pressure of 130-169 mmHg and / or a sitting clinic diastolic blood pressure of 80-109 mmHg.
* Patient has a heart rate >70 b/min at baseline (before starting bisoprolol treatment)

Exclusion Criteria:

* Secondary Hypertension
* Pregnant or lactating women and women with childbearing potential not using adequate method of contraception or agreeing to maintain sexual abstinence throughout the study;
* Unstable angina, history of myocardial infarction, stroke or coronary heart disease (coronary by-pass or angioplasty) in the previous 3 months;
* Heart failure (New York Heart Association [NYHA] III-IV);
* Haemodynamically relevant aortic or mitral valve disease;
* Obstructive hypertensive cardiomyopathy;
* Symptomatic bradycardia, second or third degree atrio-ventricular (AV) block, sick sinus syndrome, sinoatrial block, or heart rate <70 b/min at baseline (before starting bisoprolol treatment);
* Primary hyperaldosteronism;
* Renal artery stenosis;
* Impairment of hepatic or renal function as defined by liver function values of ALT ≥1.5-fold the upper normal limit or serum creatinine >150 µmol/L or upon investigator decision;
* History of intolerance to beta-blockers the drug classes used in the study.
* Patients with a known contraindication to beta-blockers, e.g. bradycardia, asthma, severe peripheral vascular disease.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Influence of the two common polymorphisms in the beta1-adrenoceptor (ADRB1) gene on changes in sitting clinic blood pressure after 6 weeks treatment with bisoprolol 2.5 mg daily. | 6 weeks
  Subjects will be divided according to the Gly389Arg and Ser49Gly polymorphisms in ADRB1 gene and the clinic blood pressure changes at 6 weeks compared between these groups.

SECONDARY OUTCOMES:
Change of blood pressure from baseline to 6 weeks by clinic sitting blood pressure according to other genotypes. | 6 weeks
  Patients will be divided into groups according to genotypes of the Fok+/Fok- polymorphism in the G-protein alpha subunit (GNAS) gene and the T393C polymorphism in the G-protein alpha subunit 1 (GNAS1) gene, and changes in blood pressure after 6 weeks treatment compared.
Change of blood pressure from baseline to 24 weeks by clinic sitting blood pressure according to other genotypes. | 24 weeks
  Patients will be divided into groups according to genotypes of the Fok+/Fok- polymorphism in the G-protein alpha subunit (GNAS) gene and the T393C polymorphism in the G-protein alpha subunit 1 (GNAS1) gene, and changes in blood pressure after 24 weeks treatment compared.
Influence of the two common polymorphisms in the beta1-adrenoceptor (ADRB1) gene on changes in ambulatory blood pressure (ABP) after 6 weeks treatment with bisoprolol 2.5 mg daily. | 6 weeks
  Subjects will be divided according to the Gly389Arg and Ser49Gly polymorphisms in the ADRB1 gene and the ambulatory blood pressure changes at 6 weeks compared between these groups.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Tomlinson, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Brian Tomlinson, Hong Kong, Hong Kong

REFERENCES:
- [Background] Hiltunen TP, Suonsyrja T, Hannila-Handelberg T, Paavonen KJ, Miettinen HE, Strandberg T, Tikkanen I, Tilvis R, Pentikainen PJ, Virolainen J, Kontula K. Predictors of antihypertensive drug responses: initial data from a placebo-controlled, randomized, cross-over study with four antihypertensive drugs (The GENRES Study). Am J Hypertens. 2007 Mar;20(3):311-8. doi: 10.1016/j.amjhyper.2006.09.006. PMID 17324745
- [Background] Suonsyrja T, Donner K, Hannila-Handelberg T, Fodstad H, Kontula K, Hiltunen TP. Common genetic variation of beta1- and beta2-adrenergic receptor and response to four classes of antihypertensive treatment. Pharmacogenet Genomics. 2010 May;20(5):342-5. doi: 10.1097/FPC.0b013e328338e1b8. PMID 20300048
- [Background] de Groote P, Helbecque N, Lamblin N, Hermant X, Mc Fadden E, Foucher-Hossein C, Amouyel P, Dallongeville J, Bauters C. Association between beta-1 and beta-2 adrenergic receptor gene polymorphisms and the response to beta-blockade in patients with stable congestive heart failure. Pharmacogenet Genomics. 2005 Mar;15(3):137-42. doi: 10.1097/01213011-200503000-00001. PMID 15861037